CLINICAL TRIAL: NCT02428517
Title: A Prospective Study Evaluating the Efficacy of the Allogeneic Hematopoietic Cell Transplantation With Antithymocyte Globulin (ATG)-Based Conditioning of Adult Acute Lymphoblastic Leukemia in First / Second Complete Hematologic Remission
Brief Title: Allogeneic Hematopoietic Cell Transplantation for Adult Acute Lymphoblastic Leukemia (2015)
Acronym: ATLAS2015
Status: Terminated | Type: Observational
Why Stopped: The PI resigned the institute, and the rest investigators at the institute decided to terminate the study.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Associate Professor, Asan Medical Center
Other Study IDs: AMC-ALLO-044
Record Dates: First submitted 2015-04-21; First posted 2015-04-28 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: acute lymphoblastic leukemia; allogeneic hematopoietic stem cell transplantation; alternative hematopoietic stem cell donor; busulfan; antithymocyte globulin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Young/MSD: Patients who are <55 years old, and will receive alloHCT for Young/MSD
  Interventions: Procedure: AlloHCT for Young/MSD
- Young/MUD&FMD: Patients who are <55 years old, and will receive alloHCT for Young/MUD&FMD
  Interventions: Procedure: AlloHCT for Young/MUD&FMD
- Old/MSD: Patients who are >=55 years old, and will receive alloHCT for Old/MSD
  Interventions: Procedure: AlloHCT for Old/MSD
- Old/MUD&FMD: Patients who are >=55 years old, and will receive alloHCT for Old/MUD&FMD
  Interventions: Procedure: AlloHCT for Old/MUD&FMD

INTERVENTIONS:
Procedure: AlloHCT for Young/MSD — Allogeneic hematopoietic cell transplantation with conditioning as follows; Busulfan 3.2 mg/kg (D-7 to D-4) Cyclophosphamide 60 mg/kg (D-3 to D-2) Thymoglobulin 1.5 mg/kg (D-3 to D-1)
  Groups: Young/MSD
Procedure: AlloHCT for Young/MUD&FMD — Allogeneic hematopoietic cell transplantation with conditioning as follows; Busulfan 3.2 mg/kg (D-7 to D-4) Fludarabine 30 mg/m2 (D-7 to D-2) Thymoglobulin 3.0 mg/kg (D-3 to D-1)
  Groups: Young/MUD&FMD
Procedure: AlloHCT for Old/MSD — Allogeneic hematopoietic cell transplantation with conditioning as follows; Busulfan 3.2 mg/kg (D-7 to D-6) Fludarabine 30 mg/m2 (D-7 to D-2) Thymoglobulin 1.5 mg/kg (D-3 to D-1)
  Groups: Old/MSD
Procedure: AlloHCT for Old/MUD&FMD — Allogeneic hematopoietic cell transplantation with conditioning as follows; Busulfan 3.2 mg/kg (D-7 to D-6) Fludarabine 30 mg/m2 (D-7 to D-2) Thymoglobulin 3.0 mg/kg (D-3 to D-1)
  Groups: Old/MUD&FMD

SUMMARY:
This study is a prospective multicenter observational study to evaluate the feasibility and the efficacy of the conditioning regimens which are modified by the donor differences and the age of recipients among patients who will receive allogeneic hematopoietic stem cell transplantation in their 1st or 2nd hematologic complete remission (CR).

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (AlloHCT) is recommended as a post-remission therapy for patients with adult ALL, and reduced intensity conditioning has been tried to decrease treatment-related mortality (TRM) rate.

Recent results showed that reduced intensity conditioning can be safely and effectively used for alloHCT of adult patients with ALL. However, the reduced intensity conditioning (RIC) can increase the possibilities of hematologic relapse, especially due to the reduced anti-leukemic effect. Another challenge in performing alloHCT for ALL is the donor availability - the limited availability of matched sibling donor (MSD) and well-matched unrelated donor (WMUD) forces us to find the feasibility of alternative donors such as partially-matched unrelated donor (PMUD) or haploidentical familial donor (familial mismatched donor, FMD).

The previous study (NCT0137764) which the investigators performed showed that the use of RIC and alternative donor was feasible. However, the incidence of relapse was slightly higher among patients who received RIC when the investigators analyzed the interim analysis results. Especially, the graft-versus-host disease (GVHD) incidence was relatively higher among patients who received alloHCT from MSD, and the investigators think that the addition of antithymocyte globulin will reduce the incidence of GVHD for these patients.

In this study, the dose of busulfan will be increased when the recipients are below 55 years old, irrespective of donor type. The investigators will also define the partially matched donor exactly and find the feasibility of PMUD and FMD again. Another endpoint for this study is to find out whether the addition of antithymocyte globulin may be helpful in preventing the GVHD incidence for patients who received alloHCT from MSD without increasing the chance of hematologic relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been previously diagnosed as one of the following disease;

  * Acute lymphoblastic leukemia
  * Biphenotypic acute leukemia with Philadelphia-positive chromosome or gene translocation
* Patients whose disease status is one of the following;

  * First hematologic complete remission (HCR1)
  * Second hematologic complete remission (HCR2)
* 15 years of age and over.
* With a suitable donor (matched sibling, well-matched unrelated, partially-matched unrelated, and haploidentical familial donor)
* Adequate cardiac function (EF>45% via cardiac scan or EchoCG)
* European Clinical Oncology Group (ECOG) performance status ≥grade 2 or Karnofsky scale >60% at the time of screening
* All patients give written informed consent according to guidelines at institution's committee on human research.

Exclusion Criteria:

* Acute lymphoblastic leukemia L3 type (Burkitt leukemia/lymphoma)
* Biphenotypic acute leukemia without BCR-ABL1 translocation
* Lymphoblastic lymphoma (bone marrow blast count is below 20% of mononuclear cells of bone marrow aspirate)
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Male patient who reject the methods of avoiding pregnancy via methods such as abstinence, barrier method (condom etc).
* Patients with a diagnosis of prior malignancy (including hematologic malignancies such as acute leukemia, lymphoma, multiple myeloma, and myelodysplastic syndrome, etc) unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed as acute lymphoblastic leukemia, who achieve hematologic complete remission for the first time or for the second time after chemotherapy, and who wil receive allogeneic hematopoietic cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
relapse-free survival (RFS) rate | 2 years
  time from achieving hematologic CR to hematologic relapse / time from the enrollment of this trial to hematologic relapse

SECONDARY OUTCOMES:
relapse-free survival (RFS) rate | 5 years
  time from achieving hematologic CR to hematologic relapse / time from the enrollment of this trial to hematologic relapse
overall survival (OS) rate | 2 years
  time from the diagnosis of disease to death/ time from the enrollment of this trial to death
overall survival (OS) rate | 5 years
  time from the diagnosis of disease to death/ time from the enrollment of this trial to death
cumulative incidence of relapse | 2 years
  from achieving hematologic CR to hematologic relapse / time from the enrollment of this trial to hematologic relapse
cumulative incidence of relapse | 5 years
  from achieving hematologic CR to hematologic relapse / time from the enrollment of this trial to hematologic relapse
treatment-related mortality rate | 100 days
  after enrollment of this trial
treatment-related mortality rate | 1 year
  after enrollment of this trial
treatment-related mortality rate | 2 years
  after enrollment of this trial
treatment-related mortality rate | 5 years
  after enrollment of this trial
cumulative incidence of acute graft-versus-host disease | 100 days
  after enrollment of this trial
cumulative incidence of acute graft-versus-host disease | 1 year
  after enrollment of this trial
cumulative incidence of acute graft-versus-host disease | 2 years
  after enrollment of this trial
cumulative incidence of acute graft-versus-host disease | 5 years
  after enrollment of this trial
cumulative incidence of chronic graft-versus-host disease | 100 days
  after enrollment of this trial
cumulative incidence of chronic graft-versus-host disease | 1 year
  after enrollment of this trial
cumulative incidence of chronic graft-versus-host disease | 2 years
  after enrollment of this trial
cumulative incidence of chronic graft-versus-host disease | 5 years
  after enrollment of this trial
molecular relapse-free survival | 2 years
  after enrollment of this trial / after achieving molecular CR (for Ph-positive ALL)

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Ma H, Sun H, Sun X. Survival improvement by decade of patients aged 0-14 years with acute lymphoblastic leukemia: a SEER analysis. Sci Rep. 2014 Feb 27;4:4227. doi: 10.1038/srep04227. PMID 24572378
- [Background] Forman SJ, Rowe JM. The myth of the second remission of acute leukemia in the adult. Blood. 2013 Feb 14;121(7):1077-82. doi: 10.1182/blood-2012-08-234492. Epub 2012 Dec 14. PMID 23243288
- [Background] Goldstone AH, Richards SM, Lazarus HM, Tallman MS, Buck G, Fielding AK, Burnett AK, Chopra R, Wiernik PH, Foroni L, Paietta E, Litzow MR, Marks DI, Durrant J, McMillan A, Franklin IM, Luger S, Ciobanu N, Rowe JM. In adults with standard-risk acute lymphoblastic leukemia, the greatest benefit is achieved from a matched sibling allogeneic transplantation in first complete remission, and an autologous transplantation is less effective than conventional consolidation/maintenance chemotherapy in all patients: final results of the International ALL Trial (MRC UKALL XII/ECOG E2993). Blood. 2008 Feb 15;111(4):1827-33. doi: 10.1182/blood-2007-10-116582. Epub 2007 Nov 29. PMID 18048644
- [Background] Bray RA, Hurley CK, Kamani NR, Woolfrey A, Muller C, Spellman S, Setterholm M, Confer DL. National marrow donor program HLA matching guidelines for unrelated adult donor hematopoietic cell transplants. Biol Blood Marrow Transplant. 2008 Sep;14(9 Suppl):45-53. doi: 10.1016/j.bbmt.2008.06.014. No abstract available. PMID 18721780
- [Background] Lee SJ, Klein J, Haagenson M, Baxter-Lowe LA, Confer DL, Eapen M, Fernandez-Vina M, Flomenberg N, Horowitz M, Hurley CK, Noreen H, Oudshoorn M, Petersdorf E, Setterholm M, Spellman S, Weisdorf D, Williams TM, Anasetti C. High-resolution donor-recipient HLA matching contributes to the success of unrelated donor marrow transplantation. Blood. 2007 Dec 15;110(13):4576-83. doi: 10.1182/blood-2007-06-097386. Epub 2007 Sep 4. PMID 17785583
- [Background] Weisdorf D, Spellman S, Haagenson M, Horowitz M, Lee S, Anasetti C, Setterholm M, Drexler R, Maiers M, King R, Confer D, Klein J. Classification of HLA-matching for retrospective analysis of unrelated donor transplantation: revised definitions to predict survival. Biol Blood Marrow Transplant. 2008 Jul;14(7):748-58. doi: 10.1016/j.bbmt.2008.04.003. PMID 18541193
- [Background] Petersdorf EW, Anasetti C, Martin PJ, Gooley T, Radich J, Malkki M, Woolfrey A, Smith A, Mickelson E, Hansen JA. Limits of HLA mismatching in unrelated hematopoietic cell transplantation. Blood. 2004 Nov 1;104(9):2976-80. doi: 10.1182/blood-2004-04-1674. Epub 2004 Jul 13. PMID 15251989
- [Background] Ballen KK, Koreth J, Chen YB, Dey BR, Spitzer TR. Selection of optimal alternative graft source: mismatched unrelated donor, umbilical cord blood, or haploidentical transplant. Blood. 2012 Mar 1;119(9):1972-80. doi: 10.1182/blood-2011-11-354563. Epub 2011 Dec 30. PMID 22210876
- [Background] Koh LP, Rizzieri DA, Chao NJ. Allogeneic hematopoietic stem cell transplant using mismatched/haploidentical donors. Biol Blood Marrow Transplant. 2007 Nov;13(11):1249-67. doi: 10.1016/j.bbmt.2007.08.003. PMID 17950913
- [Background] Reisner Y, Hagin D, Martelli MF. Haploidentical hematopoietic transplantation: current status and future perspectives. Blood. 2011 Dec 1;118(23):6006-17. doi: 10.1182/blood-2011-07-338822. Epub 2011 Sep 14. PMID 21921045
- [Background] Lee KH, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Hwang HJ, Jung AR, Kim SH, Yun SC, Shin HJ. Reduced-intensity conditioning therapy with busulfan, fludarabine, and antithymocyte globulin for HLA-haploidentical hematopoietic cell transplantation in acute leukemia and myelodysplastic syndrome. Blood. 2011 Sep 1;118(9):2609-17. doi: 10.1182/blood-2011-02-339838. Epub 2011 Jun 28. PMID 21715313
- [Background] de Lima M, Anagnostopoulos A, Munsell M, Shahjahan M, Ueno N, Ippoliti C, Andersson BS, Gajewski J, Couriel D, Cortes J, Donato M, Neumann J, Champlin R, Giralt S. Nonablative versus reduced-intensity conditioning regimens in the treatment of acute myeloid leukemia and high-risk myelodysplastic syndrome: dose is relevant for long-term disease control after allogeneic hematopoietic stem cell transplantation. Blood. 2004 Aug 1;104(3):865-72. doi: 10.1182/blood-2003-11-3750. Epub 2004 Apr 15. PMID 15090449
- [Background] Kiehl MG, Kraut L, Schwerdtfeger R, Hertenstein B, Remberger M, Kroeger N, Stelljes M, Bornhaeuser M, Martin H, Scheid C, Ganser A, Zander AR, Kienast J, Ehninger G, Hoelzer D, Diehl V, Fauser AA, Ringden O. Outcome of allogeneic hematopoietic stem-cell transplantation in adult patients with acute lymphoblastic leukemia: no difference in related compared with unrelated transplant in first complete remission. J Clin Oncol. 2004 Jul 15;22(14):2816-25. doi: 10.1200/JCO.2004.07.130. PMID 15254049
- [Background] Yakoub-Agha I, Mesnil F, Kuentz M, Boiron JM, Ifrah N, Milpied N, Chehata S, Esperou H, Vernant JP, Michallet M, Buzyn A, Gratecos N, Cahn JY, Bourhis JH, Chir Z, Raffoux C, Socie G, Golmard JL, Jouet JP; French Society of Bone Marrow Transplantation and Cell Therapy. Allogeneic marrow stem-cell transplantation from human leukocyte antigen-identical siblings versus human leukocyte antigen-allelic-matched unrelated donors (10/10) in patients with standard-risk hematologic malignancy: a prospective study from the French Society of Bone Marrow Transplantation and Cell Therapy. J Clin Oncol. 2006 Dec 20;24(36):5695-702. doi: 10.1200/JCO.2006.08.0952. Epub 2006 Nov 20. PMID 17116940
- [Background] Mohty M. Mechanisms of action of antithymocyte globulin: T-cell depletion and beyond. Leukemia. 2007 Jul;21(7):1387-94. doi: 10.1038/sj.leu.2404683. Epub 2007 Apr 5. PMID 17410187
- [Background] Baron F, Labopin M, Blaise D, Lopez-Corral L, Vigouroux S, Craddock C, Attal M, Jindra P, Goker H, Socie G, Chevallier P, Browne P, Sandstedt A, Duarte RF, Nagler A, Mohty M. Impact of in vivo T-cell depletion on outcome of AML patients in first CR given peripheral blood stem cells and reduced-intensity conditioning allo-SCT from a HLA-identical sibling donor: a report from the Acute Leukemia Working Party of the European Group for Blood and Marrow Transplantation. Bone Marrow Transplant. 2014 Mar;49(3):389-96. doi: 10.1038/bmt.2013.204. Epub 2014 Jan 13. PMID 24419525
- [Background] Dirou S, Malard F, Chambellan A, Chevallier P, Germaud P, Guillaume T, Delaunay J, Moreau P, Delasalle B, Lemarchand P, Mohty M. Stable long-term pulmonary function after fludarabine, antithymocyte globulin and i.v. BU for reduced-intensity conditioning allogeneic SCT. Bone Marrow Transplant. 2014 May;49(5):622-7. doi: 10.1038/bmt.2014.15. Epub 2014 Feb 17. PMID 24535125
- [Background] Aversa F, Tabilio A, Terenzi A, Velardi A, Falzetti F, Giannoni C, Iacucci R, Zei T, Martelli MP, Gambelunghe C, et al. Successful engraftment of T-cell-depleted haploidentical "three-loci" incompatible transplants in leukemia patients by addition of recombinant human granulocyte colony-stimulating factor-mobilized peripheral blood progenitor cells to bone marrow inoculum. Blood. 1994 Dec 1;84(11):3948-55. PMID 7524753
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Henslee-Downey PJ, Abhyankar SH, Parrish RS, Pati AR, Godder KT, Neglia WJ, Goon-Johnson KS, Geier SS, Lee CG, Gee AP. Use of partially mismatched related donors extends access to allogeneic marrow transplant. Blood. 1997 May 15;89(10):3864-72. PMID 9160695
- [Background] Kanda Y, Oshima K, Asano-Mori Y, Kandabashi K, Nakagawa M, Sakata-Yanagimoto M, Izutsu K, Hangaishi A, Tsujino S, Ogawa S, Motokura T, Chiba S, Hirai H. In vivo alemtuzumab enables haploidentical human leukocyte antigen-mismatched hematopoietic stem-cell transplantation without ex vivo graft manipulation. Transplantation. 2005 May 27;79(10):1351-7. doi: 10.1097/01.tp.0000158718.49286.14. PMID 15912103
- [Background] Huang XJ, Liu DH, Liu KY, Xu LP, Chen H, Han W, Chen YH, Wang JZ, Gao ZY, Zhang YC, Jiang Q, Shi HX, Lu DP. Haploidentical hematopoietic stem cell transplantation without in vitro T-cell depletion for the treatment of hematological malignancies. Bone Marrow Transplant. 2006 Aug;38(4):291-7. doi: 10.1038/sj.bmt.1705445. PMID 16883312
- [Background] Cho BS, Yoon JH, Shin SH, Yahng SA, Lee SE, Eom KS, Kim YJ, Lee S, Min CK, Cho SG, Kim DW, Lee JW, Min WS, Park CW, Kim HJ. Comparison of allogeneic stem cell transplantation from familial-mismatched/haploidentical donors and from unrelated donors in adults with high-risk acute myelogenous leukemia. Biol Blood Marrow Transplant. 2012 Oct;18(10):1552-63. doi: 10.1016/j.bbmt.2012.04.008. Epub 2012 Apr 16. PMID 22516055
- [Background] Rizzieri DA, Koh LP, Long GD, Gasparetto C, Sullivan KM, Horwitz M, Chute J, Smith C, Gong JZ, Lagoo A, Niedzwiecki D, Dowell JM, Waters-Pick B, Liu C, Marshall D, Vredenburgh JJ, Gockerman J, Decastro C, Moore J, Chao NJ. Partially matched, nonmyeloablative allogeneic transplantation: clinical outcomes and immune reconstitution. J Clin Oncol. 2007 Feb 20;25(6):690-7. doi: 10.1200/JCO.2006.07.0953. Epub 2007 Jan 16. PMID 17228020
- [Background] Bethge WA, Faul C, Bornhauser M, Stuhler G, Beelen DW, Lang P, Stelljes M, Vogel W, Hagele M, Handgretinger R, Kanz L. Haploidentical allogeneic hematopoietic cell transplantation in adults using CD3/CD19 depletion and reduced intensity conditioning: an update. Blood Cells Mol Dis. 2008 Jan-Feb;40(1):13-9. doi: 10.1016/j.bcmd.2007.07.001. Epub 2007 Sep 14. PMID 17869547
- [Background] Boissel N, Auclerc MF, Lheritier V, Perel Y, Thomas X, Leblanc T, Rousselot P, Cayuela JM, Gabert J, Fegueux N, Piguet C, Huguet-Rigal F, Berthou C, Boiron JM, Pautas C, Michel G, Fiere D, Leverger G, Dombret H, Baruchel A. Should adolescents with acute lymphoblastic leukemia be treated as old children or young adults? Comparison of the French FRALLE-93 and LALA-94 trials. J Clin Oncol. 2003 Mar 1;21(5):774-80. doi: 10.1200/JCO.2003.02.053. Epub 2003 Mar 1. PMID 12610173
- [Background] Nachman JB, La MK, Hunger SP, Heerema NA, Gaynon PS, Hastings C, Mattano LA Jr, Sather H, Devidas M, Freyer DR, Steinherz PG, Seibel NL. Young adults with acute lymphoblastic leukemia have an excellent outcome with chemotherapy alone and benefit from intensive postinduction treatment: a report from the children's oncology group. J Clin Oncol. 2009 Nov 1;27(31):5189-94. doi: 10.1200/JCO.2008.20.8959. Epub 2009 Oct 5. PMID 19805689
- [Background] Storring JM, Minden MD, Kao S, Gupta V, Schuh AC, Schimmer AD, Yee KW, Kamel-Reid S, Chang H, Lipton JH, Messner HA, Xu W, Brandwein JM. Treatment of adults with BCR-ABL negative acute lymphoblastic leukaemia with a modified paediatric regimen. Br J Haematol. 2009 Jun;146(1):76-85. doi: 10.1111/j.1365-2141.2009.07712.x. Epub 2009 May 4. PMID 19438471
- [Background] Mancini M, Scappaticci D, Cimino G, Nanni M, Derme V, Elia L, Tafuri A, Vignetti M, Vitale A, Cuneo A, Castoldi G, Saglio G, Pane F, Mecucci C, Camera A, Specchia G, Tedeschi A, Di Raimondo F, Fioritoni G, Fabbiano F, Marmont F, Ferrara F, Cascavilla N, Todeschini G, Nobile F, Kropp MG, Leoni P, Tabilio A, Luppi M, Annino L, Mandelli F, Foa R. A comprehensive genetic classification of adult acute lymphoblastic leukemia (ALL): analysis of the GIMEMA 0496 protocol. Blood. 2005 May 1;105(9):3434-41. doi: 10.1182/blood-2004-07-2922. Epub 2005 Jan 13. PMID 15650057
- [Background] Pullarkat V, Slovak ML, Kopecky KJ, Forman SJ, Appelbaum FR. Impact of cytogenetics on the outcome of adult acute lymphoblastic leukemia: results of Southwest Oncology Group 9400 study. Blood. 2008 Mar 1;111(5):2563-72. doi: 10.1182/blood-2007-10-116186. Epub 2007 Dec 21. PMID 18156492
- [Background] Moorman AV, Harrison CJ, Buck GA, Richards SM, Secker-Walker LM, Martineau M, Vance GH, Cherry AM, Higgins RR, Fielding AK, Foroni L, Paietta E, Tallman MS, Litzow MR, Wiernik PH, Rowe JM, Goldstone AH, Dewald GW; Adult Leukaemia Working Party, Medical Research Council/National Cancer Research Institute. Karyotype is an independent prognostic factor in adult acute lymphoblastic leukemia (ALL): analysis of cytogenetic data from patients treated on the Medical Research Council (MRC) UKALLXII/Eastern Cooperative Oncology Group (ECOG) 2993 trial. Blood. 2007 Apr 15;109(8):3189-97. doi: 10.1182/blood-2006-10-051912. Epub 2006 Dec 14. PMID 17170120
- [Background] Stock W, La M, Sanford B, Bloomfield CD, Vardiman JW, Gaynon P, Larson RA, Nachman J; Children's Cancer Group; Cancer and Leukemia Group B studies. What determines the outcomes for adolescents and young adults with acute lymphoblastic leukemia treated on cooperative group protocols? A comparison of Children's Cancer Group and Cancer and Leukemia Group B studies. Blood. 2008 Sep 1;112(5):1646-54. doi: 10.1182/blood-2008-01-130237. Epub 2008 May 23. PMID 18502832
- [Background] Thomas DA, O'Brien S, Jorgensen JL, Cortes J, Faderl S, Garcia-Manero G, Verstovsek S, Koller C, Pierce S, Huh Y, Wierda W, Keating MJ, Kantarjian HM. Prognostic significance of CD20 expression in adults with de novo precursor B-lineage acute lymphoblastic leukemia. Blood. 2009 Jun 18;113(25):6330-7. doi: 10.1182/blood-2008-04-151860. Epub 2008 Aug 14. PMID 18703706
- [Background] Chang H, Jiang A, Brandwein J. Prognostic relevance of CD20 in adult B-cell precursor acute lymphoblastic leukemia. Haematologica. 2010 Jun;95(6):1040-2; author reply 1042. doi: 10.3324/haematol.2009.021089. Epub 2010 Jan 27. No abstract available. PMID 20107157
- [Background] Campana D, Leung W. Clinical significance of minimal residual disease in patients with acute leukaemia undergoing haematopoietic stem cell transplantation. Br J Haematol. 2013 Jul;162(2):147-61. doi: 10.1111/bjh.12358. Epub 2013 May 9. PMID 23654352
- [Background] Szczepanski T. Why and how to quantify minimal residual disease in acute lymphoblastic leukemia? Leukemia. 2007 Apr;21(4):622-6. doi: 10.1038/sj.leu.2404603. Epub 2007 Feb 15. PMID 17301806